CLINICAL TRIAL: NCT06639035
Title: The Effectiveness of External Oblique Intercostal Plane Block Application in the Treatment of Acute Pain After Nephrectomy
Brief Title: The Effectiveness of External Oblique Intercostal Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Gizem Avci, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Gizem001
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative
Keywords: External Oblique Intercostal Plane Block; Nephrectomy; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Oblique Intercostal Plane Block group (Active Comparator): The External Oblique Intercostal Plane Block was administered bilaterally with local anesthetic mixture of 20 ml volume (10 ml bupivacaine 0.5%, 5 ml lidocaine 2% and 5 ml isotonic saline) after completion of surgery.
  Interventions: Other: External oblique intercostal plane block; Other: intavenous tramadol
- Control group (Placebo Comparator): At the end of the surgery, an isotonic solution was administered to the control group patients by inserting a needle through the entry site compatible with the external oblique intercostal block.
  Interventions: Other: intavenous tramadol

INTERVENTIONS:
Other: External oblique intercostal plane block — The external oblique intercostal plane block is applied to the patients at the end of the surgery.
  Arms: External Oblique Intercostal Plane Block group
Other: intavenous tramadol — Intravenous tramadol will be administered with patient-controlled analgesia

SUMMARY:
The aims of the study are as follows:To examine postoperative opioid consumption.To assess the effectiveness of external oblique intercostal plane block in managing postoperative pain in nephrectomy patients.To evaluate pain at postoperative hours 0, 2, 4, 6, 12, and 24 using the Numerical Rating Scale (NRS).To assess pain increase with movement and effort at postoperative hours 0, 2, 4, 6, 12, and 24 using NRS.

DETAILED DESCRIPTION:
The Effectiveness of External Oblique Intercostal Plane Block in the Management of Acute Pain Following NephrectomyNephrectomy is a commonly performed surgical procedure in urology due to benign or malignant reasons. Depending on the underlying pathology and the patient, the surgical procedure can vary in scale, including simple nephrectomy, partial nephrectomy, and radical nephrectomy, and may be performed either openly or laparoscopically. Postoperative pain can prolong the patient's hospital stay and impair comfort. Due to pain, patients may develop atelectasis and hypertension after surgery, leading to an increased need for narcotic analgesia. The increased demand for narcotic analgesics according to patients' age and characteristics can affect renal functions and may not improve patient comfort due to nausea and vomiting. Regional anesthesia of the torso and abdominal wall has generally focused on epidural analgesia. However, the increased use of minimally invasive laparoscopic techniques, the significance of postoperative anticoagulation regimens, and early ambulation have led to changes in analgesia selection. Although transversus abdominis plane blocks and rectus sheath blocks are frequently applied, their inability to adequately manage abdominal pain alone, along with the challenges posed in obese patients, has led to a recent shift towards the external oblique intercostal plane block.The application of the EOIP block involves the patient being in a supine position, with either the clavicle or mid-axillary line palpated to locate the 6th rib. An ultrasound probe is placed 1-2 cm lateral to the midclavicular line over the 6th rib. Under aseptic conditions, a 22-gauge 25-50 mm block needle is advanced to the 6th rib using the in-plane technique. Two ml of saline is injected for hydrodissection to ensure accurate placement. Avoiding subperiosteal injection, hydrodissection is performed between the external oblique muscle and the 6th rib. Subsequently, 20-30 ml of 0.25% bupivacaine is injected into this area. The block is then repeated on the other side.

In our clinic, a multimodal analgesia approach is preferred for patients undergoing nephrectomy. Plan blocks (administered to every suitable and consenting patient) are used in conjunction with intravenous analgesic agents. Blocks are routinely applied to patients undergoing nephrectomy, who are monitored in the postoperative intensive care unit. Our study will include suitable patients who have undergone nephrectomy and received this block. The anesthesiologist managing anesthesia will be different from the anesthetist monitoring pain. Our study is entirely observational, and no randomization will be conducted. There will be no intervention in either analgesia or anesthesia management. Patients who consent to participate will be included in the study in the recovery room after the block is administered.

The aims of the study are as follows:To examine postoperative opioid consumption.To assess the effectiveness of external oblique intercostal plane block in managing postoperative pain in nephrectomy patients.To evaluate pain at postoperative hours 0, 2, 4, 6, 12, and 24 using the Numerical Rating Scale (NRS).To assess pain increase with movement and effort at postoperative hours 0, 2, 4, 6, 12, and 24 using NRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone nephrectomy surgery.
* Aged 18-80 years
* ASA (American Society of Anesthesiologists) I-II-III risk group that underwent nephrectomy.

Exclusion Criteria:

* Patients under 18 or over 80 years of age
* Patients with a history of bleeding diathesis
* Patients with infections at the block site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours postoperatively
  All patients will receive tramadol with a patient-controlled analgesia during the postoperative period

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | 0 hours postoperatively
  NRS range will from 0- 10 with 0 being no pain and 10 the worst pain possible.
Numeric rating scale (NRS) | 2 hours postoperatively
  NRS range will from 0- 10 with 0 being no pain and 10 the worst pain possible.
Numeric rating scale (NRS) | 4 hours postoperatively
  NRS range will from 0- 10 with 0 being no pain and 10 the worst pain possible.
Numeric rating scale (NRS) | 6 hours postoperatively
  NRS range will from 0- 10 with 0 being no pain and 10 the worst pain possible.
Numeric rating scale (NRS) | 12 hours postoperatively
  NRS range will from 0- 10 with 0 being no pain and 10 the worst pain possible.
Numeric rating scale (NRS) | 24 hours postoperatively
  NRS range will from 0- 10 with 0 being no pain and 10 the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Avci, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Gizem Avcı, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. No abstract available. PMID 35249704
- [Result] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112